CLINICAL TRIAL: NCT02648113
Title: Cost-effectiveness and Cost-utility of Liberal vs Restrictive Red Blood Cell Transfusion Strategies in Patients With Acute Myocardial Infarction and Anaemia. The REALITY (REstrictive And LIberal Transfusion Strategies in Patients With Acute mYocardial Infarction) Randomized Trial.
Brief Title: Cost-effectiveness and Cost-utility of Liberal vs Restrictive Red Blood Cell Transfusion Strategies in Patients With Acute Myocardial Infarction and Anaemia.
Acronym: REALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K140705; 2015-A00360-49 (Other: ANSM)
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Myocardial Infarction; Anemia; Blood Transfusion
Keywords: Myocardial Infarction; Anemia; Blood Transfusion
MeSH Terms: conditions — Myocardial Infarction; Anemia | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restrictive transfusion strategy (Experimental): Transfusions are withheld unless Hb is <= 8 g/dL, with a target Hb of 8 to 10 g /dL
  Interventions: Procedure: Restrictive transfusion; Biological: red blood transfusion
- Liberal transfusion strategy (Experimental): Transfusions are allowed as soon as Hb <= 10 g/dL with a target of 11 g /dL.
  Interventions: Procedure: Liberal transfusion; Biological: red blood transfusion

INTERVENTIONS:
Procedure: Restrictive transfusion — Transfusions are withheld unless Hb is <= 8 g/dL, with a target Hb of 8 to 10 g /dL
  Arms: Restrictive transfusion strategy
Procedure: Liberal transfusion — transfusions are allowed as soon as Hb <= 10 g/dL with a target of 11 g /dL
  Arms: Liberal transfusion strategy
Biological: red blood transfusion

SUMMARY:
Anemia in patients with myocardial infarction (MI) is a relatively frequent issue, resulting in poorer outcome. There is equipoise regarding which transfusion strategy is best, and there is an international consensus on the urgent need for a randomized trial.

The investigators hypothesize that a "restrictive" transfusion strategy is at least non-inferior to a "liberal" transfusion strategy on 30-day outcomes of MI patients with anemia. Given the costs and risks of transfusion, a cost-effectiveness and cost-utility analysis becomes key to determining the role of each strategy.

DETAILED DESCRIPTION:
Anemia is frequent in patients with myocardial infarction (MI). The antiplatelet and anticoagulant agents used for MI treatment increase the risk of bleeding, which in turn increases the risk of ischemia and mortality. Anemia is an independent predictor of cardiac events in this setting. In the "FAST-MI 2010" nationwide registry, the prevalence of anemia (defined as Hb <10g/dL) at admission was 3% and impacted mortality. Whether this risk can be overcome by transfusion is debated.

In theory, transfusion should increase oxygen delivery to the myocardium. However, recent data suggest that oxygen delivery is not increased in patients receiving transfusion, that red blood cells are rapidly depleted of nitric oxide during storage and that, conversely, transfusion may increase platelet activation and aggregation and these consequences appear potentially even more deleterious in patients with cardiovascular disease. In the general population without cardiovascular disease of medical and surgical patients, the role of liberal vs restrictive transfusion strategies has been explored by a series of randomized trials, which have led to a consensus to withhold blood transfusions until a threshold of 7 to 8 g/dl hemoglobin is reached.

Among patients with myocardial infarction, however, both the deleterious consequences of anemia and the risks of transfusion may be greater, which leads to lingering uncertainty regarding the role of liberal vs restrictive transfusion strategies in this setting. The clinical data are observational and contradictory. Conversely, a large meta-analysis (>200 000 patients) reported a higher risk of mortality and recurrent MI in MI patients who received transfusion. More recently, a careful observational study has shown that the majority of patients undergoing blood transfusion cannot be matched with non-transfused patients due to their markedly different clinical profiles, indicating that observational studies cannot reliable establish the benefits or risks of transfusion because they are hopelessly influenced by selection bias. These results strongly highlight the need for randomized trials to establish the role of transfusion during acute MI, a call for a randomized trial that has been echoed by several thought leaders in the field in recent years. Two small randomized trials (respectively 45 and 110 patients) comparing liberal vs. restrictive transfusion strategies in MI showed no clear difference in clinical outcomes but were both underpowered.

The only guideline regarding management of anemia in this setting is from the European Society of Cardiology (ESC) guidelines on non-ST segment elevation - acute coronary syndrome (NSTE-ACS), which advise blood transfusion only if the hemodynamic status is compromised or the hemoglobin level is <7g/dL. As a result, there is wide variation in clinical practice. There is therefore equipoise regarding which transfusion strategy is best.

Hypothesis:

We hypothesize that a "restrictive" transfusion strategy (triggered by Hb <= 8 g/ dL) will be clinically non-inferior to a "liberal" transfusion strategy (triggered by Hb <= 10g/ dL) but will be less costly.

Main objective:

The main objective of the study is to compare cost-effectiveness of restrictive (triggered by Hb <= 8 g/ dL) vs liberal (triggered by Hb <= 10g/ dL) red blood transfusion strategies for patients with acute MI and anemia (7g /dL < Hb <= 10g / dL).

Secondary objective(s):

1. The key secondary objective is to perform cost-utility analyses at 30-days and 1 year.
2. The main clinical objective will be to determine whether a restrictive transfusion strategy is clinically non-inferior to a liberal transfusion strategy in terms of major adverse cardiac events (MACE) at 30 days, defined as the composite of all-cause death, nonfatal stroke, nonfatal recurrent MI, and emergency revascularization prompted by ischemia.

2. A tertiary objective will be to compare major adverse cardiac events (MACE) at 1 year, since the impact of transfusion strategies on MACE may be delayed, or conversely, an initial benefit of either strategy may become lost over the first year.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Recent acute myocardial infarction, with or without ST- segment elevation, with a combination of ischemic symptoms occurring in the past 48 hours,before the MI related admission, and elevation of biomarkers of myocardial injury (troponin)
* Anemia Hb ≤ 10g / dL but > 7 g/dL on Hb, measured at any time during the index hospital admission for MI.
* Written informed consent
* Coverage for medical insurance.

Exclusion Criteria:

* Shock (SBP < 90 mmHg with clinical signs of low output or patients requiring inotropic agents)
* MI occurring post-percutaneous coronary intervention (PCI) or post-coronary artery bypass graft (CABG) (i.e. type IV or V Acute MI according to the 2012 Universal Definition of MI
* Life-threatening or massive ongoing bleeding (as judged by the investigator)
* Any blood transfusion in the previous 30-days
* any known malignant hematologic disease Note: Sickle cell disease, thalassemia and anemia due to chronic renal failure (even under EPO) are not an exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness ratio at 30 days | 30 days
  The primary endpoint is the incremental cost-effectiveness ratio (ICER) at 30-days, using the composite endpoint (30-day composite of all-cause death, non fatal stroke, nonfatal recurrent MI, and emergency revascularization prompted by ischemia) as the effectiveness criterion

SECONDARY OUTCOMES:
Cost-effectiveness ratio at 1 year | 1 year
  Incremental cost-effectiveness ratio (ICER) at 1 year, using the composite endpoint (1-year composite of all-cause death, non fatal stroke, nonfatal recurrent MI, and emergency revascularization prompted by ischemia) as the effectiveness criterion
Clinically non inferiority at 30 days | 30 days
  The main clinical endpoint is Major Adverse Cardiac Events (MACE) at 30-days defined as the 30-day composite of all-cause death, non-fatal recurrent MI, non-fatal stroke and emergency revascularization prompted by ischemia, (all of the components of this composite clinical outcome will be analyzed separately as secondary endpoints of their own)
Clinically non inferiority at 1 year | 1 year
  The main clinical endpoint is Major Adverse Cardiac Events (MACE) at 30-days defined as the 30-day composite of all-cause death, non-fatal recurrent MI, non-fatal stroke and emergency revascularization prompted by ischemia, (all of the components of this composite clinical outcome will be analyzed separately as secondary endpoints of their own)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe-Gabriel STEG, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- Hôpital Bichat, Paris, France
- Hospital Clinic of Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Sabatine MS, Morrow DA, Giugliano RP, Burton PB, Murphy SA, McCabe CH, Gibson CM, Braunwald E. Association of hemoglobin levels with clinical outcomes in acute coronary syndromes. Circulation. 2005 Apr 26;111(16):2042-9. doi: 10.1161/01.CIR.0000162477.70955.5F. Epub 2005 Apr 11. PMID 15824203
- [Background] Hanssen M, Cottin Y, Khalife K, Hammer L, Goldstein P, Puymirat E, Mulak G, Drouet E, Pace B, Schultz E, Bataille V, Ferrieres J, Simon T, Danchin N; FAST-MI 2010 Investigators. French Registry on Acute ST-elevation and non ST-elevation Myocardial Infarction 2010. FAST-MI 2010. Heart. 2012 May;98(9):699-705. doi: 10.1136/heartjnl-2012-301700. PMID 22523054
- [Background] Silvain J, Pena A, Cayla G, Brieger D, Bellemain-Appaix A, Chastre T, Vignalou JB, Beygui F, Barthelemy O, Collet JP, Montalescot G. Impact of red blood cell transfusion on platelet activation and aggregation in healthy volunteers: results of the TRANSFUSION study. Eur Heart J. 2010 Nov;31(22):2816-21. doi: 10.1093/eurheartj/ehq209. Epub 2010 Jun 29. PMID 20591842
- [Background] Silvain J, Abtan J, Kerneis M, Martin R, Finzi J, Vignalou JB, Barthelemy O, O'Connor SA, Luyt CE, Brechot N, Mercadier A, Brugier D, Galier S, Collet JP, Chastre J, Montalescot G. Impact of red blood cell transfusion on platelet aggregation and inflammatory response in anemic coronary and noncoronary patients: the TRANSFUSION-2 study (impact of transfusion of red blood cell on platelet activation and aggregation studied with flow cytometry use and light transmission aggregometry). J Am Coll Cardiol. 2014 Apr 8;63(13):1289-1296. doi: 10.1016/j.jacc.2013.11.029. Epub 2013 Dec 18. PMID 24361322
- [Background] Yeh RW, Wimmer NJ. Blood transfusion in myocardial infarction: opening old wounds for comparative-effectiveness research. J Am Coll Cardiol. 2014 Aug 26;64(8):820-2. doi: 10.1016/j.jacc.2014.05.041. No abstract available. PMID 25145527
- [Background] Carson JL, Grossman BJ, Kleinman S, Tinmouth AT, Marques MB, Fung MK, Holcomb JB, Illoh O, Kaplan LJ, Katz LM, Rao SV, Roback JD, Shander A, Tobian AA, Weinstein R, Swinton McLaughlin LG, Djulbegovic B; Clinical Transfusion Medicine Committee of the AABB. Red blood cell transfusion: a clinical practice guideline from the AABB*. Ann Intern Med. 2012 Jul 3;157(1):49-58. doi: 10.7326/0003-4819-157-1-201206190-00429. PMID 22751760
- [Background] Carson JL, Carless PA, Hebert PC. Outcomes using lower vs higher hemoglobin thresholds for red blood cell transfusion. JAMA. 2013 Jan 2;309(1):83-4. doi: 10.1001/jama.2012.50429. PMID 23280228
- [Background] Wu WC, Rathore SS, Wang Y, Radford MJ, Krumholz HM. Blood transfusion in elderly patients with acute myocardial infarction. N Engl J Med. 2001 Oct 25;345(17):1230-6. doi: 10.1056/NEJMoa010615. PMID 11680442
- [Background] Chatterjee S, Wetterslev J, Sharma A, Lichstein E, Mukherjee D. Association of blood transfusion with increased mortality in myocardial infarction: a meta-analysis and diversity-adjusted study sequential analysis. JAMA Intern Med. 2013 Jan 28;173(2):132-9. doi: 10.1001/2013.jamainternmed.1001. PMID 23266500
- [Background] Salisbury AC, Reid KJ, Marso SP, Amin AP, Alexander KP, Wang TY, Spertus JA, Kosiborod M. Blood transfusion during acute myocardial infarction: association with mortality and variability across hospitals. J Am Coll Cardiol. 2014 Aug 26;64(8):811-9. doi: 10.1016/j.jacc.2014.05.040. PMID 25145526
- [Background] Rao SV, Sherwood MW. Isn't it about time we learned how to use blood transfusion in patients with ischemic heart disease? J Am Coll Cardiol. 2014 Apr 8;63(13):1297-1299. doi: 10.1016/j.jacc.2013.11.028. Epub 2013 Dec 18. No abstract available. PMID 24361316
- [Background] Cooper HA, Rao SV, Greenberg MD, Rumsey MP, McKenzie M, Alcorn KW, Panza JA. Conservative versus liberal red cell transfusion in acute myocardial infarction (the CRIT Randomized Pilot Study). Am J Cardiol. 2011 Oct 15;108(8):1108-11. doi: 10.1016/j.amjcard.2011.06.014. Epub 2011 Jul 24. PMID 21791325
- [Background] Carson JL, Brooks MM, Abbott JD, Chaitman B, Kelsey SF, Triulzi DJ, Srinivas V, Menegus MA, Marroquin OC, Rao SV, Noveck H, Passano E, Hardison RM, Smitherman T, Vagaonescu T, Wimmer NJ, Williams DO. Liberal versus restrictive transfusion thresholds for patients with symptomatic coronary artery disease. Am Heart J. 2013 Jun;165(6):964-971.e1. doi: 10.1016/j.ahj.2013.03.001. Epub 2013 Apr 8. PMID 23708168
- [Background] Hamm CW, Bassand JP, Agewall S, Bax J, Boersma E, Bueno H, Caso P, Dudek D, Gielen S, Huber K, Ohman M, Petrie MC, Sonntag F, Uva MS, Storey RF, Wijns W, Zahger D; ESC Committee for Practice Guidelines. ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: The Task Force for the management of acute coronary syndromes (ACS) in patients presenting without persistent ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2011 Dec;32(23):2999-3054. doi: 10.1093/eurheartj/ehr236. Epub 2011 Aug 26. No abstract available. PMID 21873419
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Hebert PC, Yetisir E, Martin C, Blajchman MA, Wells G, Marshall J, Tweeddale M, Pagliarello G, Schweitzer I; Transfusion Requirements in Critical Care Investigators for the Canadian Critical Care Trials Group. Is a low transfusion threshold safe in critically ill patients with cardiovascular diseases? Crit Care Med. 2001 Feb;29(2):227-34. doi: 10.1097/00003246-200102000-00001. PMID 11246298
- [Background] Villanueva C, Colomo A, Bosch A, Concepcion M, Hernandez-Gea V, Aracil C, Graupera I, Poca M, Alvarez-Urturi C, Gordillo J, Guarner-Argente C, Santalo M, Muniz E, Guarner C. Transfusion strategies for acute upper gastrointestinal bleeding. N Engl J Med. 2013 Jan 3;368(1):11-21. doi: 10.1056/NEJMoa1211801. PMID 23281973
- [Background] Sherwood MW, Rao SV. Acute coronary syndromes: Blood transfusion in patients with acute MI and anaemia. Nat Rev Cardiol. 2013 Apr;10(4):186-7. doi: 10.1038/nrcardio.2013.14. Epub 2013 Feb 5. PMID 23380974
- [Background] Perkins HA, Busch MP. Transfusion-associated infections: 50 years of relentless challenges and remarkable progress. Transfusion. 2010 Oct;50(10):2080-99. doi: 10.1111/j.1537-2995.2010.02851.x. No abstract available. PMID 20738828
- [Background] Williamson LM, Devine DV. Challenges in the management of the blood supply. Lancet. 2013 May 25;381(9880):1866-75. doi: 10.1016/S0140-6736(13)60631-5. PMID 23706803
- [Background] Bernard AC, Davenport DL, Chang PK, Vaughan TB, Zwischenberger JB. Intraoperative transfusion of 1 U to 2 U packed red blood cells is associated with increased 30-day mortality, surgical-site infection, pneumonia, and sepsis in general surgery patients. J Am Coll Surg. 2009 May;208(5):931-7, 937.e1-2; discussion 938-9. doi: 10.1016/j.jamcollsurg.2008.11.019. Epub 2009 Mar 26. PMID 19476865
- [Background] Vincent JL, Baron JF, Reinhart K, Gattinoni L, Thijs L, Webb A, Meier-Hellmann A, Nollet G, Peres-Bota D; ABC (Anemia and Blood Transfusion in Critical Care) Investigators. Anemia and blood transfusion in critically ill patients. JAMA. 2002 Sep 25;288(12):1499-507. doi: 10.1001/jama.288.12.1499. PMID 12243637
- [Background] Frank SM, Abazyan B, Ono M, Hogue CW, Cohen DB, Berkowitz DE, Ness PM, Barodka VM. Decreased erythrocyte deformability after transfusion and the effects of erythrocyte storage duration. Anesth Analg. 2013 May;116(5):975-981. doi: 10.1213/ANE.0b013e31828843e6. Epub 2013 Feb 28. PMID 23449853
- [Background] Vamvakas EC, Blajchman MA. Transfusion-related mortality: the ongoing risks of allogeneic blood transfusion and the available strategies for their prevention. Blood. 2009 Apr 9;113(15):3406-17. doi: 10.1182/blood-2008-10-167643. Epub 2009 Feb 2. PMID 19188662
- [Background] Murray CJ, Richards MA, Newton JN, Fenton KA, Anderson HR, Atkinson C, Bennett D, Bernabe E, Blencowe H, Bourne R, Braithwaite T, Brayne C, Bruce NG, Brugha TS, Burney P, Dherani M, Dolk H, Edmond K, Ezzati M, Flaxman AD, Fleming TD, Freedman G, Gunnell D, Hay RJ, Hutchings SJ, Ohno SL, Lozano R, Lyons RA, Marcenes W, Naghavi M, Newton CR, Pearce N, Pope D, Rushton L, Salomon JA, Shibuya K, Vos T, Wang H, Williams HC, Woolf AD, Lopez AD, Davis A. UK health performance: findings of the Global Burden of Disease Study 2010. Lancet. 2013 Mar 23;381(9871):997-1020. doi: 10.1016/S0140-6736(13)60355-4. Epub 2013 Mar 5. PMID 23668584
- [Background] Husereau D, Drummond M, Petrou S, Carswell C, Moher D, Greenberg D, Augustovski F, Briggs AH, Mauskopf J, Loder E; CHEERS Task Force. Consolidated Health Economic Evaluation Reporting Standards (CHEERS) statement. BMJ. 2013 Mar 25;346:f1049. doi: 10.1136/bmj.f1049. PMID 23529982
- [Background] Briggs AH, O'Brien BJ. The death of cost-minimization analysis? Health Econ. 2001 Mar;10(2):179-84. doi: 10.1002/hec.584. PMID 11252048
- [Background] Kaiser C, Brunner-La Rocca HP, Buser PT, Bonetti PO, Osswald S, Linka A, Bernheim A, Zutter A, Zellweger M, Grize L, Pfisterer ME; BASKET Investigators. Incremental cost-effectiveness of drug-eluting stents compared with a third-generation bare-metal stent in a real-world setting: randomised Basel Stent Kosten Effektivitats Trial (BASKET). Lancet. 2005 Sep 10-16;366(9489):921-9. doi: 10.1016/S0140-6736(05)67221-2. PMID 16154019
- [Background] Caruba T, Katsahian S, Schramm C, Charles Nelson A, Durieux P, Begue D, Juilliere Y, Dubourg O, Danchin N, Sabatier B. Treatment for stable coronary artery disease: a network meta-analysis of cost-effectiveness studies. PLoS One. 2014 Jun 4;9(6):e98371. doi: 10.1371/journal.pone.0098371. eCollection 2014. PMID 24896266
- [Background] Greiner W, Weijnen T, Nieuwenhuizen M, Oppe S, Badia X, Busschbach J, Buxton M, Dolan P, Kind P, Krabbe P, Ohinmaa A, Parkin D, Roset M, Sintonen H, Tsuchiya A, de Charro F. A single European currency for EQ-5D health states. Results from a six-country study. Eur J Health Econ. 2003 Sep;4(3):222-31. doi: 10.1007/s10198-003-0182-5. PMID 15609189
- [Background] Fearon WF, Shilane D, Pijls NH, Boothroyd DB, Tonino PA, Barbato E, Juni P, De Bruyne B, Hlatky MA; Fractional Flow Reserve Versus Angiography for Multivessel Evaluation 2 (FAME 2) Investigators. Cost-effectiveness of percutaneous coronary intervention in patients with stable coronary artery disease and abnormal fractional flow reserve. Circulation. 2013 Sep 17;128(12):1335-40. doi: 10.1161/CIRCULATIONAHA.113.003059. Epub 2013 Aug 14. PMID 23946263
- [Background] Wijeysundera HC, Tomlinson G, Ko DT, Dzavik V, Krahn MD. Medical therapy v. PCI in stable coronary artery disease: a cost-effectiveness analysis. Med Decis Making. 2013 Oct;33(7):891-905. doi: 10.1177/0272989X13497262. Epub 2013 Jul 25. PMID 23886676
- [Background] Magnuson EA, Farkouh ME, Fuster V, Wang K, Vilain K, Li H, Appelwick J, Muratov V, Sleeper LA, Boineau R, Abdallah M, Cohen DJ; FREEDOM Trial Investigators. Cost-effectiveness of percutaneous coronary intervention with drug eluting stents versus bypass surgery for patients with diabetes mellitus and multivessel coronary artery disease: results from the FREEDOM trial. Circulation. 2013 Feb 19;127(7):820-31. doi: 10.1161/CIRCULATIONAHA.112.147488. Epub 2012 Dec 31. PMID 23277307
- [Background] Raikou M, Briggs A, Gray A, McGuire A. Centre-specific or average unit costs in multi-centre studies? Some theory and simulation. Health Econ. 2000 Apr;9(3):191-8. doi: 10.1002/(sici)1099-1050(200004)9:33.0.co;2-1. PMID 10790698
- [Background] Hollingworth W, McKell-Redwood D, Hampson L, Metcalfe C. Cost-utility analysis conducted alongside randomized controlled trials: are economic end points considered in sample size calculations and does it matter? Clin Trials. 2013 Feb;10(1):43-53. doi: 10.1177/1740774512465358. Epub 2012 Dec 11. PMID 23231969
- [Background] Mauskopf JA, Sullivan SD, Annemans L, Caro J, Mullins CD, Nuijten M, Orlewska E, Watkins J, Trueman P. Principles of good practice for budget impact analysis: report of the ISPOR Task Force on good research practices--budget impact analysis. Value Health. 2007 Sep-Oct;10(5):336-47. doi: 10.1111/j.1524-4733.2007.00187.x. PMID 17888098
- [Background] Robinson SD, Janssen C, Fretz EB, Berry B, Chase AJ, Siega AD, Carere RG, Fung A, Simkus G, Klinke WP, Hilton JD. Red blood cell storage duration and mortality in patients undergoing percutaneous coronary intervention. Am Heart J. 2010 May;159(5):876-81. doi: 10.1016/j.ahj.2010.02.018. PMID 20435199
- [Result] Ducrocq G, Gonzalez-Juanatey JR, Puymirat E, Lemesle G, Cachanado M, Durand-Zaleski I, Arnaiz JA, Martinez-Selles M, Silvain J, Ariza-Sole A, Ferrari E, Calvo G, Danchin N, Avendano-Sola C, Frenkiel J, Rousseau A, Vicaut E, Simon T, Steg PG; REALITY Investigators. Effect of a Restrictive vs Liberal Blood Transfusion Strategy on Major Cardiovascular Events Among Patients With Acute Myocardial Infarction and Anemia: The REALITY Randomized Clinical Trial. JAMA. 2021 Feb 9;325(6):552-560. doi: 10.1001/jama.2021.0135. PMID 33560322
- [Result] Ducrocq G, Calvo G, Gonzalez-Juanatey JR, Durand-Zaleski I, Avendano-Sola C, Puymirat E, Lemesle G, Arnaiz JA, Martinez-Selles M, Rousseau A, Cachanado M, Vicaut E, Silvain J, Karam C, Danchin N, Simon T, Steg PG; REALITY investigators. Restrictive vs liberal red blood cell transfusion strategies in patients with acute myocardial infarction and anemia: Rationale and design of the REALITY trial. Clin Cardiol. 2021 Feb;44(2):143-150. doi: 10.1002/clc.23453. Epub 2021 Jan 6. PMID 33405291
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066
- [Derived] Ducrocq G, Cachanado M, Simon T, Puymirat E, Lemesle G, Lattuca B, Ariza-Sole A, Silvain J, Ferrari E, Gonzalez-Juanatey JR, Martinez-Selles M, Lermusier T, Coste P, Vanzetto G, Cottin Y, Dillinger JG, Calvo G, Steg PG; REALITY Investigators. Restrictive vs Liberal Blood Transfusions for Patients With Acute Myocardial Infarction and Anemia by Heart Failure Status: An RCT Subgroup Analysis. Can J Cardiol. 2024 Sep;40(9):1705-1714. doi: 10.1016/j.cjca.2024.02.013. Epub 2024 Feb 24. PMID 38408702
- [Derived] Durand-Zaleski I, Ducrocq G, Mimouni M, Frenkiel J, Avendano-Sola C, Gonzalez-Juanatey JR, Ferrari E, Lemesle G, Puymirat E, Berard L, Cachanado M, Arnaiz JA, Martinez-Selles M, Silvain J, Ariza-Sole A, Calvo G, Danchin N, Paco S, Drouet E, Abergel H, Rousseau A, Simon T, Steg PG. Economic evaluation of restrictive vs. liberal transfusion strategy following acute myocardial infarction (REALITY): trial-based cost-effectiveness and cost-utility analyses. Eur Heart J Qual Care Clin Outcomes. 2023 Feb 28;9(2):194-202. doi: 10.1093/ehjqcco/qcac029. PMID 35612990
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836